CLINICAL TRIAL: NCT05502224
Title: Pilot Project for the Implementation of an Integrated Multidisciplinary Follow-up for Young Patients With Breast Cancer or Germ Cell Tumor
Brief Title: Multidisciplinary Approach to Fatigue
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IJB-PRINTEMPS-2022
Record Dates: First submitted 2022-08-11; First posted 2022-08-16 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer; Germ Cell Tumor
MeSH Terms: conditions — Breast Neoplasms; Neoplasms, Germ Cell and Embryonal

STUDY DESIGN:
Intervention Model Description: Each individual is his own control. It is therefore a longitudinal data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Specific fatigue management program (Other)
  Interventions: Other: Ergospirometry

INTERVENTIONS:
Other: Ergospirometry — Maximum aerobic capacity (VO2 max), Maximum load, Ventilatory threshold and the patient's RQ

SUMMARY:
Prospective longitudinal, single-center, non-randomized study for the implementation of an integrated multidisciplinary fatigue follow-up for young patients with breast cancer or germ cell tumour

DETAILED DESCRIPTION:
Each patient will receive a full evaluation by a multidisciplinary evaluation by a multidisciplinary team during one day. This evaluation will take place between 1 and 3 months after the end of "acute" treatments. The team is composed of an oncologist, a psychologist, a physiotherapist, a dietician and a nurse-coach. The goal of this comprehensive evaluation is to :

* to detect organic or psychological factors (severe depression,...) contributing to fatigue.
* to evaluate in detail the impact of fatigue on the patient's daily life.
* to evaluate the patient's level of physical activity in order to propose an adequate and and personalized management. During this evaluation, the patient will be asked to discuss which aspects of his or her daily life he or she would like to improve as a priority. At the end of this complete evaluation, each patient's case will be will be discussed in a multidisciplinary meeting with all the people involved in the program in order to propose a detailed and personalized treatment plan.

This plan will be explained in detail to the patient by the nurse-coach who will organize and coordinate the patient's care. The patient will receive the detailed management plan in writing.

The patient will receive the detailed management plan in writing, which will also be communicated to the patient's treating physicians.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 39 years at the time of signing the informed consent
* Patient who speaks and understands French
* Signed study informed consent form obtained prior to any study related procedures
* At minimum, a moderate (>3) fatigue level according to the Standard Rating Scale (NRS) 1 month after completion of acute treatment; as measured at the Survivorship of the standard program
* Patient with either: curative breast cancer (AJCC stage I-II-III) or a germ cell tumor

Exclusion Criteria:

* Refusal to participate in the study
* Patient having chosen to participate in another psychosocial intervention study for the duration of the study.
* Patients with AJCC stage IV breast cancer

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-19 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Evaluate the feasibility of the specific fatigue management program | Through study completion, an average of 4 years
  Rate of participation The program will be considered feasible for a given patient if he/she participates in a minimum of 70% of the 70% of the sessions/activities defined in their particular program

SECONDARY OUTCOMES:
The measurement of the evolution of the intensity of residual fatigue in the months following acute cancer treatment(s) before and after the specific fatigue management program | At the time of multidisciplinary screening and at 1, 3, 6, 12 and 18 months after completion of the specific fatigue management program.
  Numerical Rating Scale (NRS) for fatigue

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Jules Bordet, Brussels, Belgium